CLINICAL TRIAL: NCT04342832
Title: CRyoballoon Ablation Versus mediCal thErapy in Patients With Heart Failure and Atrial Fibrillation: A Multicenter Randomized Clinical Trial, the RACE-8-HF Trial
Brief Title: Cryoballoon Ablation Versus Medical Therapy in Patients With Heart Failure and Atrial Fibrillation
Acronym: RACE-8-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment speed
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL71710.068.19
Record Dates: First submitted 2020-03-26; First posted 2020-04-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure, Systolic
Keywords: Pulmonary vein isolation; Cryoballoon ablation; Atrial fibrillation; Heart failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: Multicenter randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early invasive treatment (cryoballoon ablation) (Active Comparator)
  Interventions: Procedure: Cryoballoon ablation
- Standard medical care (No Intervention)

INTERVENTIONS:
Procedure: Cryoballoon ablation — If a patient is randomized to early invasive treatment, the ablation is performed within 3 months by an experienced cardiac electrophysiologist using CE-certified equipment. Via the femoral vein a guiding catheter is advanced through the inferior vena cava to the right atrium and into the left atrium via transseptal puncture. Then, the cryoballoon is advanced, inflated, and placed against one of the four PVs. PV occlusion is assessed by selective contrast injection. When adequate PV antral seal is confirmed, ablation of the tissue in contact with the balloon is performed using pressurized liquid nitrous oxide. The cold inflated balloon thus creates circular lesions around the PV. The balloon and tissue interface are then allowed to reach normal temperatures. Depending on local practice, the freeze-thaw cycle may be repeated twice. Electrical isolation is assessed and when it is confirmed, the next PV is treated in the same way. The procedure ends when all PV's are isolated.
  Other Names: Pulmonary vein isolation; PVI; CBA
  Arms: Early invasive treatment (cryoballoon ablation)

SUMMARY:
Rationale:

Atrial fibrillation (AF) and heart failure (HF) can cause each other and sustain each other. Combined, the two diseases negatively influence each other's prognosis and lead to higher mortality. Studies in HF patients in which the AF burden is reduced by AF ablation show promising results toward improved prognosis, but so far only one randomized trial is conducted that focused on major clinical endpoints. As the selected patients in this trial were not representative for the entire population and its ablation method varied from patient to patient, it is the aim of the present study to confirm that early invasive therapy consisting of a strict pulmonary vein isolation (PVI) protocol using cryoballoon therapy has positive effects on hard clinical endpoints in a wider variety of patients in the HF population.

Furthermore, there are no studies which compare cost-effectiveness of an early invasive strategy in this patient category. The investigators expect that avoided hospitalizations and healthcare resource utilizations lead to lower costs in the AF ablation group, despite initial higher costs of the procedure.

Objective:

To compare outcome and cost-effectiveness of early AF ablation by PVI using cryoballoon therapy with standard (medical) therapy in patients with heart failure with reduced ejection fraction.

Study design:

Multicenter, randomized, open label clinical trial.

Study population:

Symptomatic adult patients with heart failure with reduced ejection fraction (<40%) and paroxysmal or persistent AF.

Intervention:

AF ablation (PVI) using cryoballoon therapy.

Outcome measures:

The primary endpoint is a combined endpoint of all-cause mortality, unplanned cardiovascular hospitalization, and stroke (time-to-event analysis).

Secondary endpoints of the trial are:

* A combined endpoint of mortality, number of unplanned cardiovascular hospitalizations, and stroke (recurrent-event analysis);
* A hierarchical endpoint of mortality, unplanned cardiovascular hospitalizations, stroke, and HF complaints;
* Cost-effectiveness. Key exploratory endpoints include individual components of the combined endpoints, days alive out of the hospital, hospitalizations for heart failure, recurrence of atrial arrhythmia, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80;
* HF with ejection fraction <40%, as assessed by recent (<6 months) echocardiography or cardiovascular magnetic resonance imaging (CMR);
* AF, documented on standard ECG or Holter monitoring;
* Eligible for both treatment arms;
* Signed and dated informed consent prior to admission to the trial.

Exclusion Criteria:

* End-stage heart failure: NYHA class IV, patients on waiting list for cardiac transplant and/or left ventricular assist device;
* Long-standing (> 1 year) persistent or permanent AF;
* Previous pulmonary vein isolation or surgical ablation;
* Left atrial diameter ≥60 mm or left atrial volume index ≥50 ml/m2;
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) ≤25 ml/min/1.73m2;
* Recent (<90 days) acute coronary syndrome, cardiac intervention1, or stroke/transient ischemic attack (TIA);
* Planned or expected cardiac surgery in the following year;
* Active infectious disease or malignancy;
* Women who are pregnant or planning to become pregnant during the trial;
* Contraindication for cryoballoon ablation or other condition that may prevent subjects from adhering to the trial protocol, in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, unplanned cardiovascular hospitalizations and stroke (time-to-event analysis) | Study duration (1-5 years, expected median follow-up duration 2 years)

SECONDARY OUTCOMES:
Combined endpoint of all-cause mortality | Study duration (1-5 years, expected median follow-up duration 2 years)
Total number of unplanned cardiovascular hospitalizations and stroke (recurrent-event analysis) | Study duration (1-5 years, expected median follow-up duration 2 years)
Hierarchal endpoint of all-cause mortality, unplanned cardiovascular hospitalizations, stroke and change in heart failure complaints (hierarchical endpoint analysis) | Study duration (1-5 years, expected median follow-up duration 2 years)
Cost-effectiveness | Study duration (1-5 years, expected median follow-up duration 2 years)
Budget impact | Study duration (1-5 years, expected median follow-up duration 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Vernooy, MD PhD, Study Chair — Maastricht UMC+, Radboudumc; Michiel Rienstra, MD PhD, Study Chair — UMC Groningen
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No